CLINICAL TRIAL: NCT05604573
Title: DNA Mutation Detection in Circulating Tumor DNA and Tissue by Massive Multiplex Allele Discrimination Priming System(mmADPS) for Pancreatic Cancer
Brief Title: DNA Mutation Detection in Circulating Tumor DNA and Tissue by mmADPS for Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: GENECAST Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Other Study IDs: H-2111-047-1271
Record Dates: First submitted 2022-10-24; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Circulating Tumor DNA; DNA mutation; DNA methylation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection; Mutation; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pancreatic cancer: patients with pancreatic cancer
  Interventions: Diagnostic Test: cell free DNA in blood, genetic mutation in tissue
- control: patients without any malignancy
  Interventions: Diagnostic Test: cell free DNA in blood, genetic mutation in tissue

INTERVENTIONS:
Diagnostic Test: cell free DNA in blood, genetic mutation in tissue — Diagnostic test for cell free DNA in blood, genetic mutation in tissue

SUMMARY:
Based on the cell free nucleic acid analysis information of blood samples and genetic mutation profile of EUS-FNB tissue from pancreatic cancer, the concordance between them is evaluated. And based on this information, biomarkers for diagnosis, treatment, and prognosis of pancreatic cancer are explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer through histological or radiologic examination and before treatment begins
* Patients aged 18 or older who voluntarily agrees to participate in the study and is willing to understand and comply with the subsequent treatment procedures and sample collection schedule
* Among patients diagnosed with benign pancreatic diseases (pancreatic cyst, chronic pancreatitis, etc.), patients who have need for histological examination as control group

Exclusion Criteria:

* Where the subject himself/herself refuses to fill out the consent form or is unable to fill out the consent form
* If a laboratory test is impossible due to a qualitative problem with the collected blood sample
* Where the collected tissue does not contain tissue of the desired malignant or benign disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or older who diagnosed with pancreatic cancer through histological or radiologic examination and before treatment begins
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
correlation of genetic mutation | the day of study enrollment (baseline)
  concordance of genetic mutation between tissue and blood of treatment-naive status
detection sensitivity of genetic mutation by mmADPS | the day of study enrollment (baseline)
  detection sensitivity of genetic mutation by mmADPS

SECONDARY OUTCOMES:
correlation of genetic mutation and prognosis | through study completion, an average of 1 year
  correlation of genetic mutation and prognosis

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea